CLINICAL TRIAL: NCT06158555
Title: Targeted Perfusion Based Haemodynamic Management in Critically Ill Patients Using Urethral Perfusion - a Pilot Study
Brief Title: Targeted Perfusion Based Haemodynamic Management in Critically Ill Patients Using Urethral Perfusion
Acronym: TARGET UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 315717
Record Dates: First submitted 2023-08-31; First posted 2023-12-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Patients will receive fluid and vasopressor challenges and the macro and microvascular responses will be recorded using the IKORUS monitor alongside conventional haemodynamic monitoring
  Interventions: Drug: 250 ML NaCl 4.5 MG/ML Injection

INTERVENTIONS:
Drug: 250 ML NaCl 4.5 MG/ML Injection — Bolus 250 ml crystalloid. Usually 0.9% saline or compound sodium lactate solution at discretion of attending clinician

SUMMARY:
To assess the safety and feasibility of the IKORUS device in critically ill patients and to gather exploratory data on haemodynamic coherence

ELIGIBILITY:
Inclusion Criteria:

* Within 24 h of ICU admission
* Predicted length of ICU stay at least 5 days
* Receiving >0.1 mcg/kg/min of noradrenaline at time of study enrolment

Exclusion Criteria:

* Palliative treatment intent
* Contra indication to urethral catheterisation or complication during previous urethral catheter insertion
* Contraindication to fluid or vasopressor challenges in the opinion of the attending clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change to Urethral Perfusion Index | 5 minutes after fluid challenge administration

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No